CLINICAL TRIAL: NCT06058325
Title: Healthy School Lunch at Primary Schools in Rotterdam, the Netherlands
Brief Title: Healthy School Lunches at Primary Schools in Rotterdam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Wilma Jansen, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 10115
Record Dates: First submitted 2023-08-31; First posted 2023-09-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: Healthy lunch; Diet; Children; School; Effectivity; Feasibility

STUDY DESIGN:
Intervention Model Description: The investigators will use a cross-over design, which means participating schools have both a control and intervention period during academic year 2023-2024. Schools will be randomized into group A or B, starting with either an intervention or control period.
  During the intervention period, schools will organize a healthy lunch for all children during four days a week for a duration of half an academic year (approximately 18 weeks). During the control period, children will bring their own lunch box.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Students will bring their own lunch box in the control period.
- Intervention group (Experimental): Students will get a healthy lunch at school in the intervention period.
  Interventions: Other: Healthy school lunch

INTERVENTIONS:
Other: Healthy school lunch — The healthy school lunch will be co-created together with school staff, parents, and children, and should be healthy according guidelines of the Dutch nutrition center.
  Arms: Intervention group

SUMMARY:
Obesity in children is increasing over the last decades and the majority of children in Europe fails to have a healthy diet. In the Netherlands, the majority of primary schools do not provide a (healthy) school lunch. However, previous research shows some positive effects. Within the current study the investigators want to implement healthy school lunches in the city of Rotterdam, a city with a very diverse youth population. The main objective of the healthy school lunch project is to evaluate the effectiveness and feasibility of providing healthy school lunches.

This is a prospective, single center, intervention study using a cross-over design with 3 measurement moments to collect data on effects and feasibility. Additional feasibility data will be collected throughout the study via questionnaires for teachers.

The study population is derived from primary schools participating in the "Enjoy Being Fit!" program in the city of Rotterdam. Children (4-12 years old) from these schools are eligible to participate in this study. Children from participating primary schools will take part in observations and complete questionnaires (only grade 5 to 8). Parents and teachers will complete questionnaires.

Together with individual schools and stakeholders a healthy school-lunch concept will be developed and implemented for half a school year. Data will be collected on three time points during the school year.

Questionnaires for children and parents will focus on dietary behaviour/food intake, taste preferences, perceived health, and the satisfaction with the healthy school lunch (also for teachers). Atmosphere in the class during lessons and during lunch will be measured in questionnaires for children and teachers. The questionnaire for parents also focuses on affordability of a healthy school lunch. Observation forms will be used to score on one day what snack and lunch children bring to/get at school.

ELIGIBILITY:
Inclusion Criteria:

* Schools: Schools will be included if they are a LF! school, have a high deprivation score and ≥ 20% overweight/obesity, and are willing to participate in the project irrespective of starting in the intervention or control period. Schools should be willing to facilitate retrieving consent from parents and should provide students time to complete the questionnaire during school hours. They should also be willing to participate in a co-creation event, in which the lunch concept for their school will be designed together with school staff, parents, and children. Schools should be willing to facilitate the implementation of a healthy school lunch and should not provide any extra activities regarding healthy school lunches during the control period.
* Children: All children of the participating schools will be eligible to receive a healthy school lunch, also if parents do not provide informed consent for the research project. Data will be gathered for all children for whom informed consent is provided for participating in the data gathering. Informed consent must be signed by the parents of children who are allowed to participate in the research activities (observations and questionnaires) in the school. Additionally, when children are 12 years or older they have to sign an informed consent themselves.
* Parents: All parents with children in the participating schools will be included into the project to complete questionnaires. Informed consent must be signed by the parent.
* Teachers: All teachers in participating will be included into the project to complete questionnaires. Informed consent must be signed by the teacher.

Exclusion Criteria:

* The non-compliance of the inclusion criteria will be considered as exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Dietary content of children's lunches - assessed by an observation form | Three times during academic year 2023-2024: baseline/approximately 18 weeks/approximately 36 weeks
  Observation of type and amount of bread, topping, drinks, fruits, vegetables, and other food products

SECONDARY OUTCOMES:
General dietary behaviour of children - assessed by a questionnaire | Three times during academic year 2023-2024: baseline/approximately 18 weeks/approximately 36 weeks
  (consumption of breakfast, fruit, vegetable, water, sugar sweetened beverages -children and parents)
  Questions adapted from the GGD (Dutch municipal health service) health monitor.
Perceived health of children - assessed by a questionnaire | Three times during academic year 2023-2024: baseline/approximately 18 weeks/approximately 36 weeks
  Questions adapted from the GGD (Dutch municipal health service) health monitor: general health, in past week, in past 3 months.
Taste preferences of children - assessed by a questionnaire | Three times during academic year 2023-2024: baseline/approximately 18 weeks/approximately 36 weeks
  Self-reported questions on taste of different fruits (n=12) and vegetables (n=16).
  Questions adapted from the Healthy Primary School of the Future study
Concentration in class - assessed by a questionnaire | Three times during academic year 2023-2024: baseline/approximately 18 weeks/approximately 36 weeks
  Self-reported question on the ability to concentrate in class. For children reported on individual level. For teachers reported on class level.
Atmosphere in class - assessed by a questionnaire | Three times during academic year 2023-2024: baseline/approximately 18 weeks/approximately 36 weeks
  Self-reported questions on the atmosphere in class. For children reported on individual level. For teachers reported on class level.
Financial situation of parents - assessed by a questionnaire | During intervention arm: depending on the group either approximately 18 weeks after baseline or approximately 36 weeks after baseline
  Questions adapted from the GGD (Dutch municipal health service) health monitor: difficulties making ends meet & inability to do things due to lack of money
Satisfaction of the healthy school lunch - assessed by a questionnaire | During intervention arm: depending on the group either approximately 18 weeks after baseline or approximately 36 weeks after baseline
  Self-reported questions partly adapted from the Healthy School Lunch study and partly constructed by the research team. Satisfaction questions focused on: participation, content of lunch, organization, reasons to participate, continuation.
  Descriptives will be presented.

OTHER OUTCOMES:
Demographic variables - assessed by a questionnaire | Three times during academic year 2023-2024: baseline/approximately 18 weeks/approximately 36 weeks
  age, gender, country of birth
Type of dietary requirement(s) - assessed by a questionnaire | Three times during academic year 2023-2024: baseline/approximately 18 weeks/approximately 36 weeks
  The kind and amount of dietary requirements will be collected by using a self-reported question.
  Descriptives will be presented.
Feasibility data on implementation and sustainability - assessed by a questionnaire | Every month during academic year 2023-2024: baseline/1 month/2 months/ 3 months/ 4 months/ 5 months/ 6 months/ 7 months/ 8 months/ 9 months
  Feasibility data on implementation and sustainability will be collected via self-reported questions constructed by the research team. Questions will focus on implementation, organization, time investment, sustainability.
  Open answers will be analyzed qualitatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health, Erasmus MC University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
A data sharing statement will be finalized when known which percentage of participants consent for sharing data outside of our own organization.

REFERENCES:
- [Background] Hahnraths MTH, Willeboordse M, van Assema P, Winkens B, van Schayck CP. The Effects of the Healthy Primary School of the Future on Children's Fruit and Vegetable Preferences, Familiarity and Intake. Nutrients. 2021 Sep 17;13(9):3241. doi: 10.3390/nu13093241. PMID 34579117
- [Background] van Kleef E, Rongen FC, Vingerhoeds MH, Dijkstra SC, Seidell JC. Improving dietary intake during lunch through the provision of a healthy school lunch at Dutch primary schools: design of a pretest-posttest effectiveness study. BMC Public Health. 2020 May 12;20(1):662. doi: 10.1186/s12889-020-08807-1. PMID 32398052
- [Derived] Wargers A, Polychronakis K, Nieboer D, Raat H, Jansen W. Co-creation and implementation of a healthy lunch at Dutch primary schools in disadvantaged neighbourhoods: design of a cluster randomised cross-over effectiveness study. BMJ Open. 2024 Oct 16;14(10):e083534. doi: 10.1136/bmjopen-2023-083534. PMID 39414278